CLINICAL TRIAL: NCT01698697
Title: A Single Centre, Randomized, Balanced Double-blind, Cross-Over Trial Investigating the Bioequivalence of a Continuous Subcutaneous Infusion of a Marketed NovoRapid Formulation Containing 100 U/ml and a New NovoRapid Formulation Containing 200 U/ml in Healthy Male Volunteers
Brief Title: Comparison of Two Insulin Aspart Formulations in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NN248-1494
Record Dates: First submitted 2012-09-28; First posted 2012-10-03 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2017-02

CONDITIONS: Diabetes; Healthy
MeSH Terms: conditions — Diabetes Mellitus | interventions — Insulin Aspart

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- U100 (Active Comparator)
  Interventions: Drug: insulin aspart
- U200 (Experimental)
  Interventions: Drug: insulin aspart

INTERVENTIONS:
Drug: insulin aspart — Bolus 0.1 U/kg administered simultaneously with a continuous infusion of 0.029 U/kg/h via a programmed insulin pump. A total dose of 0.35 U/kg is delivered to the subject in the 12 hour infusion

SUMMARY:
This trial is conducted in Africa. The aim of this trial is to determine if a new formulation (U200) of insulin aspart containing 200 U/mL is bioequivalent to that of a marketed insulin aspart formulation (U100).

ELIGIBILITY:
Inclusion Criteria:

* Normal findings in medical history and physical examination unless the investigator considers any abnormality to be clinically irrelevant
* Normal laboratory values, electrocardiogram (ECG), and vital signs unless the investigator considers any abnormality to be clinically irrelevant
* Body mass index (BMI) 18-26 kg/m^2 (both inclusive)
* Weight 60-90 kg
* Non-smoker

Exclusion Criteria:

* Any condition requiring the regular use of any medication
* Known or suspected allergy to the trial product or related products
* Family history of type 1 diabetes mellitus

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2002-09-02 (Actual); Primary Completion 2002-10-18 (Actual); Study Completion 2002-10-18 (Actual)

PRIMARY OUTCOMES:
Area under the curve (AUC)
Area under the glucose infusion rate curve

SECONDARY OUTCOMES:
Cmax (maximum plasma concentration)
Time to reach maximum (tmax)
Terminal half-life (t½)
Incidence of hypoglycemic events
Adverse events
GIRmax: The maximal GIR (glucose infusion rate)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Bloemfontein, South Africa

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com